CLINICAL TRIAL: NCT00981201
Title: A Randomized, Double-Blind Study of the Biological Effects and Tolerability of Celecoxib as a Chemopreventive Agent in Current and Former Smokers
Brief Title: Celecoxib as a Chemopreventive Agent in Current and Former Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ID00-230
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2009-09

CONDITIONS: Smoking; Prevention
Keywords: Smoking; Cancer Prevention; Celecoxib; Celebrex; Placebo
MeSH Terms: conditions — Smoking | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Celecoxib + Placebo (Experimental)
  Interventions: Drug: Celecoxib; Drug: Placebo
- Celecoxib + Celecoxib (Experimental)
  Interventions: Drug: Celecoxib
- Placebo + Celecoxib (Active Comparator)
  Interventions: Drug: Celecoxib; Drug: Placebo
- Placebo + Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Months 1-3:
  As of October, 2003, the starting dose for celecoxib will be 400 mg by mouth twice daily. (Note: Prior to October, 2003, the starting dose for celecoxib was 200 mg by mouth twice daily.)
  Other Names: Celebrex
  Arms: Celecoxib + Celecoxib; Celecoxib + Placebo
Drug: Celecoxib — Months 4-6:
  As of October, 2003, the starting dose for celecoxib will be 400 mg by mouth twice daily. (Note: Prior to October, 2003, the starting dose for celecoxib was 200 mg by mouth twice daily.)
  Other Names: Celebrex
  Arms: Celecoxib + Celecoxib; Placebo + Celecoxib
Drug: Placebo — Months 1-3:
  By mouth twice daily.
  Arms: Placebo + Celecoxib; Placebo + Placebo
Drug: Placebo — Months 4-6:
  By mouth twice daily.
  Arms: Celecoxib + Placebo; Placebo + Placebo

SUMMARY:
The purpose of this study is:

* To examine the effect of celecoxib treatment on Ki-67 expression, a marker of cell proliferation, in the bronchial epithelium of current and former smokers.
* To examine the toxicity associated with celecoxib administration.
* To measure the effect of celecoxib treatment on arachidonic acid metabolites in the bronchial epithelium of current and former smokers.

DETAILED DESCRIPTION:
COX-2 is an enzyme thought to be involved in the development of some cancer. Celecoxib is a COX-2 inhibitor.

Before treatment begins, participants will have a bronchoscopy (tissue sample from the lung). This is taken to see if different elements (biomarkers) in the tissue can predict which individuals are at higher risk for developing cancer. In a bronchoscopy a tube will be placed through the nose into the lung (while under sedation) to remove tissue samples for laboratory analysis (biopsy). Cells will also be collected during the bronchoscopy by spraying the lungs with a small amount water and then removing the water (bronchial lavage, bronchial washing). In addition, a sputum sample will be taken and the inside of the cheek will be scraped (buccal sample).

A complete physical exam will be performed before beginning treatment and at 1, 2, 3, 4, 5, and 6 months. During these visits, participants will be asked questions about tobacco/alcohol exposure. Participants will have blood taken before beginning treatment and at 1, 3, 4, and 6 months. Urine samples will be taken before beginning treatment and at 3 and 6 months. The research nurse will also ask participants about any adverse signs or symptoms that they have experienced. Participants who smoke will be encouraged to stop smoking. Sources for assistance to stop smoking will be provided for all study participants who continue to smoke.

In this study, participants will be randomly picked (as in the toss of a coin) to be in one of four treatment groups. Treatment in this study will last 6 months. Participants in the first group will receive a placebo during all 6 months. A placebo is a substance that looks like the study drug but is inactive. Participants in the second group will receive a placebo during Months 1-3 and Celecoxib during Months 4-6. Participants in the third group will receive Celecoxib during Months 1-3 and placebo during Months 4-6. Participants in the fourth group will receive Celecoxib during all 6 months. Neither the participant nor the participant's doctor will know to which treatment group the participant was assigned. Participants have an equal chance of being assigned to any of these groups.

Participants will take 2 capsules twice a day for the 6-month treatment period. The capsule could be either a placebo or the study drug.

At 3 and 6 months, participants will have a physical exam, blood tests, and a bronchoscopy. Participants should take their study medication with a sip of water 2 hours before each bronchoscopy with a sip of water. Sputum and buccal samples will also be taken at these times. The research nurse will ask participants questions about changes and/or additions to the medications.

This is an investigational study. The use of Celecoxib in the prevention of lung cancer is investigational. Up to 250 individuals will take part in this study. All will be enrolled at the M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18-74 years old.
2. Participants must have at least a 20 pack-year history of smoking.
3. Participants may have had a prior laryngeal cancer (Stage I or II) that was completely resected or rendered disease-free by radiation therapy, or a prior lung cancer (Stage I NSCLC) that was completely resected, without radiotherapy. Participants must have been clinically free of any cancer for at least 6 months.
4. Participants must have no contraindications for undergoing bronchoscopy.
5. Participants must have no active pulmonary infections.
6. Participants must not be taking inhaled steroids or oral non-steroidal anti-inflammatory drugs on a regular basis. (Low dose aspirin <= 81 mg/day is allowed.)
7. Participants must have the following blood levels: total granulocyte count > 1500; platelet count > 100,000; total bilirubin <= 1.5 mg %; and creatinine <= 1.5 mg %.
8. Participants must complete the pretreatment evaluation and must consent to bronchoscopy and to endobronchial biopsy for documentation of histologic status.
9. Participants must sign a study-specific informed consent form.

Exclusion Criteria:

1. Participants with active gastric or duodenal ulcers or a history of ulcers requiring prophylactic H2 blockers.
2. Participants with active pulmonary infections or recent history of pulmonary infection (within 1 month).
3. Participants receiving inhaled steroid therapy on a regular basis.
4. Participants with acute intercurrent illness, or participants who had surgery within the preceding 4 weeks unless they have fully recovered.
5. Participants requiring chronic ongoing treatment with NSAIDs.
6. Participants who are allergic to aspirin or sulfanamides.
7. Participants with history of stroke, transient ischemic attack, uncontrolled hypertension, and/or angina pectoris.
8. Participants who are pregnant and/or breast-feeding.
9. Participants (men or women) of childbearing potential who are not using an effective method of contraception.
10. History of cardiovascular diseases that might include one of the following: myocardial infarction, angina, coronary angioplasty, congestive heart failure, stroke, or coronary bypass surgery.
11. Diagnosis of diabetes
12. History of deep venous thrombosis, pulmonary embolism, systemic lupus erythematous, family history of protein S or C deficiencies, prior heparin-induced thrombocytopenia, or known Factor V Leiden mutation.
13. Family history of premature CAD. This is defined as individuals with either: 1) father with MI prior to age 55, or 2) mother with MI prior to age 60.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2001-11; Primary Completion 2007-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The change of the proliferation marker Ki-67. | From baseline to 3-month visit.

SECONDARY OUTCOMES:
The changes in tissue COX-2 expression, lavage PGE2 levels, and genetic markers such as LOH, chromosome instability, and chromosome polysomy. | 3-months and 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M. Kurie, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States